CLINICAL TRIAL: NCT00553670
Title: Predictor and Mechanism of a Side Branch Jail After Main Branch Stent Implantation in Bifurcation Lesions
Brief Title: Mechanism and Predictor of Side Branch Jailing
Acronym: PRESSURE
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Other Study IDs: H-0707-022-212
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Bifurcating Coronary Artery Lesions; Main Branch Stent Implantation; Side Branch Jailing
Keywords: coronary artery; bifurcation; stent; intravascular ultrasound; fractional flow reserve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients with elective coronary intervention for LAD-diagonal bifurcation lesion with provisional side branch intervention strategy with successful intravascular ultrasound and fractional flow reserve measurement

SUMMARY:
Coronary artery bifurcation lesion is still one of the most challenging lesion subsets in the field of non-surgical treatment for a stenotic coronary artery. When one stent is placed in the main brach, it increases the side branch's stenosis degree. However, its mechanism and incidence are not known. This study will be performed to search for the mechanism and incidence of that phenomenon.

ELIGIBILITY:
Inclusion Criteria:

1. Elective coronary intervention (including stabilized ACS patients)
2. Bifurcation lesion with TIMI 3 flow
3. Side branch diameter > 2mm, side branch lesion length < 10mm by visual estimation

Exclusion Criteria:

1. Left main coronary disease
2. AMI, or Old MI at LAD territory
3. LVEF < 40%, or other significant valvular or myocardial disease
4. Significant side branch distal lesion
5. Angiographically visible thrombus
6. Heavily calcified lesion
7. Side branch predilatation before main branch stent implantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bifurcating coronary artery lesion in left anterior descending coronary artery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Koo BK, Waseda K, Kang HJ, Kim HS, Nam CW, Hur SH, Kim JS, Choi D, Jang Y, Hahn JY, Gwon HC, Yoon MH, Tahk SJ, Chung WY, Cho YS, Choi DJ, Hasegawa T, Kataoka T, Oh SJ, Honda Y, Fitzgerald PJ, Fearon WF. Anatomic and functional evaluation of bifurcation lesions undergoing percutaneous coronary intervention. Circ Cardiovasc Interv. 2010 Apr;3(2):113-9. doi: 10.1161/CIRCINTERVENTIONS.109.887406. PMID 20407111